CLINICAL TRIAL: NCT04525235
Title: The Effect of High Dose Rifampicin on the Activity of Cytochrome P450 Enzymes and P-glycoprotein in Patients With Pulmonary Tuberculosis: a Cocktail Phenotyping Study
Brief Title: Phenotyping of High Dose Rifampicin
Acronym: PHENORIF
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: PHENORIF
Record Dates: First submitted 2020-08-20; First posted 2020-08-25 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — Digoxin; Caffeine; Tolbutamide; Midazolam; Dextromethorphan; Omeprazole; Rifampin

STUDY DESIGN:
Intervention Model Description: each participants will receive phenotyping probe drugs with the standard dose of rifampicin and with a high dose rifampicin in a fixed oreder
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rifampicin standard dose (Active Comparator): rifampicin standard dose + phenotyping cocktail
  Interventions: Combination Product: phenotyping cocktail; Drug: rifampicin
- Rifampicin high dose (Experimental): rifampicin high dose + phenotyping cocktail
  Interventions: Combination Product: phenotyping cocktail; Drug: rifampicin

INTERVENTIONS:
Combination Product: phenotyping cocktail — A single dose of a cocktail of phenotyping probe drugs (caffeine, tolbutamide, omeprazole, dextromethorphan, midazolam and digoxin) will be administered together with standard dose rifampicin and 40 mg/kg rifampicin, respectively. Blood samples will be taken to assess phenotyping metrics of the cocktail agents and rifampicin pharmacokinetic parameters. The effect of high and standard dose rifampicin on the phenotyping metrics of the cocktail agents will be compared by using the bioequivalence approach
  Other Names: digoxin; caffeine; tolbutamide; midazolam; dextromethorphan; omeprazole
Drug: rifampicin — A single dose of a cocktail of phenotyping probe drugs (caffeine, tolbutamide, omeprazole, dextromethorphan, midazolam and digoxin) will be administered together with standard dose rifampicin and 40 mg/kg rifampicin, respectively. Blood samples will be taken to assess phenotyping metrics of the cocktail agents and rifampicin pharmacokinetic parameters. The effect of high and standard dose rifampicin on the phenotyping metrics of the cocktail agents will be compared by using the bioequivalence approach

SUMMARY:
Higher doses of rifampicin as a means of more efficient use of this pivotal TB drug has shown promising results and might become standard in future. This means that higher doses of rifampicin will be co-administered with many other drugs taken by TB patients, including anti-retroviral, anti-diabetic, cardiovascular and other drugs. Therefore, in this study the aim is to quantitatively assess the drug interaction potential of high dose rifampicin (~40 mg/kg daily dose, the currently available maximum tolerated dose) with respect to five major human drug-metabolizing CYP enzymes and P-gp in comparison to the conventional dose of 10 mg/kg daily in pulmonary TB patients. A phenotyping approach with single administration of several selective substrates for multiple enzymes will be used, in order to prevent multiple drug-drug interaction studies.

ELIGIBILITY:
Inclusion Criteria:

* The participant is able and willing to provide written, informed consent prior to all trial-related procedures.
* The participant is aged between 18 and 65 years, inclusive.
* The participant is a diagnosed pulmonary TB patient.
* The participant is currently being treated with a daily dose of 10 mg/kg rifampicin, i.e. 450 mg daily for patients with a body weight below 55 kg and 600 mg daily for participants with a body weight above 55 kg. This is in correspondence with the local South African TB treatment programme. Furthermore, the participant has to be in the continuation phase of the treatment regimen (i.e. month 3 to 6), has demonstrated reasonable treatment compliance (≥80% of doses) and tolerates treatment well.
* The participant has a body weight (in light clothing and with no shoes) between 40 and 85 kg, inclusive.
* The participant is and stays non-pregnant (based on a negative serum pregnancy test,) and non-lactating (female participants of childbearing potential only).

Exclusion Criteria:

* The patient is in poor general condition where any change in treatment cannot be accepted per discretion of the Investigator.
* The participant has active Hepatitis B.
* The participant has active Hepatitis C.
* The participant is receiving antiretroviral therapy (ART).
* There is evidence showing the participant has clinically significant metabolic, gastrointestinal, or other abnormalities than could possibly alter the PK of rifampicin and/or the probe drugs.
* The participant has a history of or current clinically relevant cardiovascular disorder such as:
* heart failure, atrioventricular (AV) block, arrhythmia, tachyarrhythmia or status after myocardial infarction.
* family history of sudden death of unknown or cardiac-related cause, or of prolonged QTc interval.
* The participant has clinically relevant abnormalities in the ECG such as atrioventricular (AV) block, prolongation of the QRS complex over 100 milliseconds, or of a QTc interval over 450 milliseconds on the screening ECG.
* The participant has abnormal alanine aminotransferase (ALT) and/or aspartate transferase (AST) levels > 3 times the upper limit of the laboratory reference range at screening.
* The participant has a known or suspected, current drug or amphetamine abuse, that is, in the opinion of the Investigator, sufficient to compromise the safety or cooperation of the patient.
* The participant used any drugs or substances known to be strong inhibitors or inducers of cytochrome P450 enzymes and/or P-glycoprotein (P-gp) within 2 weeks prior to day 1 (i.e. 1 month before administration of the phenotyping probes on day 15) of the study (including carbamazepine, barbiturates, St. John's Wort, clarithromycin, itraconazole, fluconazole, quinidine, ketoconazole, erythromycin). Exceptions may be made for participants who have received 3 days or less of one of these drugs or substances, if there has been a wash-out period equivalent to at least 5 half-lives of that drug or substance before day 1 of the study.
* The participant uses any of the phenotyping probe drugs (i.e. midazolam, caffeine, dextromethorphan, tolbutamide, omeprazole and digoxin) as part of standard medical treatment.
* The participant has as history of allergy to any of the phenotyping probe drugs (i.e. midazolam, caffeine, dextromethorphan, tolbutamide, omeprazole and digoxin).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-01-07 (Actual); Primary Completion 2021-08-12 (Actual); Study Completion 2021-08-12 (Actual)

PRIMARY OUTCOMES:
area under the curve | 24 hours
  area under the curve of probe drugs

CONTACTS AND LOCATIONS:
Locations (2):
- South Africa (2):
  - TASK, Cape Town
  - UCT lung institute, Cape Town

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stemkens R, Jager Vd, Dawson R, Diacon AH, Narunsky K, Padayachee SD, Boeree MJ, van Beek SW, Colbers A, Coenen MJH, Svensson EM, Fuhr U, Phillips PPJ, Te Brake LHM, Aarnoutse RE; PanACEA consortium. Drug interaction potential of high-dose rifampicin in patients with pulmonary tuberculosis. Antimicrob Agents Chemother. 2023 Oct 18;67(10):e0068323. doi: 10.1128/aac.00683-23. Epub 2023 Sep 28. PMID 37768317